CLINICAL TRIAL: NCT02026271
Title: A Phase I Study of Ad-RTS-hIL-12, an Inducible Adenoviral Vector Engineered to Express hIL-12 in the Presence of the Activator Ligand Veledimex in Subjects With Recurrent or Progressive Glioblastoma or Grade III Malignant Glioma
Brief Title: A Study of Ad-RTS-hIL-12 With Veledimex in Subjects With Glioblastoma or Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-102
Record Dates: First submitted 2013-12-16; First posted 2014-01-01 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma Multiforme; Anaplastic Oligoastrocytoma
MeSH Terms: conditions — Glioblastoma | interventions — veledimex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad-RTS-hIL-12+veledimex (Experimental): varying doses of intratumoral Ad-RTS-hIL-12 (INXN-2001) and oral veledimex (activator ligand).
  Interventions: Biological: Ad-RTS-hIL-12; Drug: veledimex

INTERVENTIONS:
Biological: Ad-RTS-hIL-12 — * 2.0 x 10^11 viral particles (vp) per injection or 1.0 x 10^12 viral particles (vp) per injection
  * one intratumoral injection of Ad-RTS-hIL-12
  Other Names: INXN-2001
Drug: veledimex — * 4 doses (20mg/day, 40mg/day, 80mg/day, and 120mg/day)
  * 14 oral daily doses of veledimex
  * 1 Expansion cohort at a single dose level at or below MTD
  Other Names: INXN-1001; Activator Ligand

SUMMARY:
This research study involves an investigational product: Ad-RTS-hIL-12 given with veledimex for production of human IL-12. IL-12 is a protein that can improve the body's natural response to disease by enhancing the ability of the immune system to kill tumor cells and may interfere with blood flow to the tumor.

The main purpose of this study is to evaluate the safety and tolerability of a single tumor injection of Ad-RTS-hIL-12 given with oral veledimex.

DETAILED DESCRIPTION:
Eligible patients will be stratified to one of two groups, according to clinical indication for tumor resection. Patients who are scheduled for a standard of care craniotomy and tumor resection will receive one dose of veledimex before the resection procedure. Ad-RTS-hIL-12 will be administered by free-hand injection. Patients will continue on oral veledimex for 14 days.

Patients not scheduled for tumor resection will receive Ad-RTS-hIL-12 by stereotactic injection and then will continue on oral veledimex for 14 days.

The study is divided into three periods: the screening period, the treatment period and the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 and ≤ 75 years of age
2. Provision of written informed consent for tumor resection, stereotactic surgery, tumor biopsy, samples collection and treatment with investigational products prior to undergoing any study procedures
3. Histologically confirmed supratentorial glioblastoma or other WHO grade III or IV malignant glioma from archival tissue.
4. Evidence of tumor recurrence/progression by MRI (RANO criteria) post standard initial therapy.
5. Previous standard of care anti-tumor treatment including surgery and/or biopsy and chemoradiation. The washout periods from prior therapies are intended as follows:

   1. Nitrosoureas: 6 weeks
   2. Other cytotoxic agents: 4 weeks
   3. Anti-angiogenic agents including bevacizumab: 4 weeks
   4. Targeted agents including small-molecule tyrosine kinase inhibitors: 2 weeks
   5. Experimental immunotherapies: 3 months
   6. Vaccine based therapy: 3 months
6. Able to undergo standard MRI scans with contrast agent
7. Karnofsky Performance Status ≥ 70
8. Adequate bone marrow reserves and liver and kidney function, as assessed by the following laboratory requirements:

   1. Hemoglobin ≥ 9 g/L
   2. Lymphocytes > 500/ mm3
   3. Absolute Neutrophil Count ≥ 1500/ mm3
   4. Platelets ≥ 100,000/ mm3
   5. Serum creatinine ≤ 1.5 x ULN
   6. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN. For subjects with documented liver metastases, ALT and AST ≤ 5 × ULN
   7. Total bilirubin < 1.5 x ULN
   8. International Normalized Ratio (INR) and activated Partial Thromboplastin Time [PTT] within normal institutional limits
9. Male and female subjects must agree to use a highly reliable method of birth control (expected failure rate less than 5% per year) from the screening visit through 28 days after the last dose of study drug. Women of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Radiotherapy within 4 weeks or less prior to starting first veledimex dose
2. Subjects with clinically significant increased intracranial pressure or uncontrolled seizures.
3. Known immunosuppressive disease, autoimmune conditions, and /or chronic viral infections
4. Use of systemic antibacterials, antifungals or antivirals for the treatment of acute clinically significant infection within 2 weeks of first veledimex dose. Concomitant therapy for chronic infections is not allowed. Subjects must be afebrile prior to Ad-RTS-hIL-12 injection; only prophylactic antibiotic use is permitted perioperatively.
5. Use of enzyme-inducing anti-epileptic drugs (EIAED) within 7 days prior to the first dose of study drug.
6. Other concurrent clinically active malignant disease, requiring treatment, with the exception of non-melanoma cancers of the skin or carcinoma in-situ of the cervix or non-metastatic prostate cancer.
7. Nursing or pregnant females
8. Prior exposure to veledimex
9. Use of medications that induce, inhibit or are substrates of CYP450 3A4 within 7 days prior to the first veledimex dosing
10. Presence of any contra-indication for a neurosurgical procedure
11. Unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator or medical monitor, jeopardize the safety of a subject and/or their compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (6):
- United States (6):
  - Cedars-Sinai, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Northwestern, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Brigham & Women's, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Chiocca EA, Yu JS, Lukas RV, Solomon IH, Ligon KL, Nakashima H, Triggs DA, Reardon DA, Wen P, Stopa BM, Naik A, Rudnick J, Hu JL, Kumthekar P, Yamini B, Buck JY, Demars N, Barrett JA, Gelb AB, Zhou J, Lebel F, Cooper LJN. Regulatable interleukin-12 gene therapy in patients with recurrent high-grade glioma: Results of a phase 1 trial. Sci Transl Med. 2019 Aug 14;11(505):eaaw5680. doi: 10.1126/scitranslmed.aaw5680. PMID 31413142

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Plan: 4 Veledimex (V) doses (20, 40, 80, 120 mg QD) and 2 AdRTShIL12 doses (2x10^11vp, 1x10^12vp).
  Actual: V 10, 20, 30, 40 mg and AdRTShIL12 2x10^11vp. Grp 1: After 20mg cohort, SRC approved 40mg which was deemed the MAD due to DLTs. SRC approved 30mg cohort to determine MTD, but due to compliance SRC opened a 20mg exp cohort then inter 10mg cohort. Based on V compliance and OS, 20mg was determined as the optimal dose.
  Grp 2: Spnsr decided not to escalate post Cohort 1 (not safety based).
Groups:
- Group 1 (Intracranial) 10 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 10 mg/day 3 (± 2) hours before the craniotomy procedure. Immediately after tumor resection, subjects will receive Ad-RTS-hIL-12 2 x 10^11 vp and then will continue on oral veledimex for 14 days.
- Group 1 (Intracranial) 20 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 20 mg/day 3 (± 2) hours before the craniotomy procedure. . Immediately after tumor resection, subjects will receive Ad-RTS-hIL-12 2 x 10^11 vp and then will continue on oral veledimex for 14 days.
- Group 1 (Intracranial) 30 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 30 mg/day 3 (± 2) hours before the craniotomy procedure. Immediately after tumor resection, subjects will receive Ad-RTS-hIL-12 2 x 10^11 vp and then will continue on oral veledimex for 14 days.
- Group 1 (Intracranial) 40 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 40 mg/day 3 (± 2) hours before the craniotomy procedure. Immediately after tumor resection, subjects will receive Ad-RTS-hIL-12 2 x 10^11 vp and then will continue on oral veledimex for 14 days.
- Group 2 (Stereotactic) 20 mg/Day Veledimex: Subjects who will not undergo tumor resection will receive Ad-RTS-hIL-12 (2 x 10^11) by standard stereotactic surgery on Day 0. After the Ad-RTS-hIL-12 injection, veledimex 20 mg/day will be administered orally for 14 days.
Period: Overall Study
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Started | 6 | 16 | 4 | 6 | 8
Enrolled | 6 | 16 | 4 | 6 | 8
Treated | 6 | 16 | 4 | 6 | 7
Overall Safety Population (OSP) | 6 | 16 | 4 | 6 | 7
Evaluable Safety Population (ESP) | 6 | 15 | 4 | 6 | 7
Pharmacokinetic Population (PKP) | 6 | 15 | 4 | 6 | 7
Completed | 4 | 13 | 2 | 3 | 7
Not Completed | 2 | 3 | 2 | 3 | 1
Not completed — Adverse Event | 2 | 3 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS): Overall Safety Population (OSP) includes all subjects who have received at least one dose of veledimex (pretumor resection and) and/or all subjects who received Ad-RTS-hIL-12. The FAS will be used for summaries of baseline characteristics and safety.
Groups:
- Group 1 (Intracranial) 10 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 10 mg/day 3 (± 2) hours before the craniotomy procedure.
- Group 1 (Intracranial) 20 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 20 mg/day 3 (± 2) hours before the craniotomy procedure.
- Group 1 (Intracranial) 30 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 30 mg/day 3 (± 2) hours before the craniotomy procedure.
- Group 1 (Intracranial) 40 mg/Day Veledimex: Group 1: Subjects scheduled for craniotomy and tumor resection: Subjects with a clinical indication for tumor resection will receive veledimex 40 mg/day 3 (± 2) hours before the craniotomy procedure.
- Group 2 (Stereotactic) 20 mg/Day Veledimex: Subjects who will not undergo tumor resection will receive Ad-RTS-hIL-12 by standard stereotactic surgery on Day 0. After the Ad-RTS-hIL-12 injection, veledimex 20 mg/day will be administered orally for 14 days.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex | Total
Number analyzed (Participants) | 6 | 16 | 4 | 6 | 7 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.87 (12.39) | 46.90 (13.22) | 60.40 (15.12) | 48.12 (9.32) | 51.71 (17.16) | 49.64 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 2 | 4 | 5 | 25
  Male | 3 | 5 | 2 | 2 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 6 | 15 | 3 | 6 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2
  White | 5 | 15 | 4 | 6 | 6 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 4 | 6 | 7 | 39
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 172.75 (9.92) | 174.69 (8.75) | 169.53 (15.96) | 176.08 (12.11) | 175.64 (7.16) | 174.25 (9.71)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 79.86 (9.10) | 81.11 (18.78) | 73.70 (25.99) | 86.84 (20.26) | 83.66 (6.22) | 81.49 (16.61)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Varying Doses of Intratumoral Ad-RTS-hIL-12 and Oral Veledimex Doses in Subjects With Recurrent or Progressive Glioblastoma or Grade III Malignant Glioma
Description: Evaluation will be based on the incidence, intensity, and type of Adverse Events (AEs). Clinically significant changes in the subjects' physical examinations, vital signs, and ECG evaluations, and clinical manifestations relevant to abnormal laboratory values will be captured as AEs.
Time Frame: 3 years
Population: The Full Analysis Set (FAS): Overall Safety Population (OSP) includes all subjects who have received at least one dose of veledimex (pretumor resection and) and/or all subjects who received Ad-RTS-hIL-12.
Measure: Number; unit: participants
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 6 | 16 | 4 | 6 | 7
participants
  Any TEAEs | 6 | 16 | 4 | 5 | 7
  Any Serious TEAEs | 2 | 10 | 3 | 4 | 4
  Any TEAEs with Toxicity Grade ≥ 3 | 4 | 11 | 4 | 5 | 4
  Any TEAEs Leading to Treatment Dose Modification | 3 | 4 | 2 | 2 | 2
  Any TEAEs Leading to Treatment Discontinuations | 2 | 3 | 2 | 3 | 0
  Any TEAEs Leading to Death | 1 | 2 | 1 | 0 | 3
  Any Drug-Related TEAEs | 6 | 10 | 4 | 5 | 4
  Any Drug-Related Serious TEAEs | 1 | 7 | 2 | 3 | 2
  Any Drug-Related TEAEs with Toxicity Grade ≥ 3 | 4 | 6 | 2 | 4 | 2
  Any Drug-Related TEAEs Leading to Treatment Dose Modification | 3 | 4 | 2 | 2 | 2
  Any Drug-Related TEAEs Leading to Treatment Discontinuations | 2 | 2 | 2 | 3 | 0
  Any Drug-Related TEAEs Leading to Death | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Veledimex Maximum Tolerated Dose (MTD) When Given With Varying Doses of Intratumoral Ad-RTS-hIL-12
Description: The protocol defined the MTD as the dose level below at which less than 33% of subjects, of the same cohort in a group, experienced DLTs, with an independent assessment of Group 1 and Group 2 subjects.
  • The number of DLTs and the proportion of subjects with any DLT and each type of DLT were summarized by veledimex dose within each group.
Time Frame: 3 years
Population: •The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP was used for analysis of DLTs.
Measure: Number; unit: participants
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 6 | 15 | 4 | 6 | 7
participants
  Total participants with DLTs | 2 | 4 | 0 | 3 | 0
  DLT of Alanine Aminotransferase Increased | 2 | 0 | 0 | 0 | 0
  DLT of Leukopenia | 0 | 1 | 0 | 0 | 0
  DLT of Thrombocytopenia | 0 | 1 | 0 | 0 | 0
  DLT of Meningitis Aseptic | 0 | 1 | 0 | 0 | 0
  DLT of Liver Function Test Increased | 0 | 1 | 0 | 0 | 0
  DLT of Cytokine Release Syndrome | 0 | 0 | 0 | 2 | 0
  DLT of Aspartate Aminotransferase Increased | 0 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Group 1 (Intracranial) 10 mg/Day Veledimex vs Group 1 (Intracranial) 20 mg/Day Veledimex vs Group 1 (Intracranial) 30 mg/Day Veledimex vs Group 1 (Intracranial) 40 mg/Day Veledimex; Test type: Other; MTD was not determined in this study. Dose escalation decision rules were based on a standard 3+3 design modified to independently evaluate the two stratified subject groups that may exhibit different safety and tolerability profiles. The study was planned to explore 4 veledimex (V) dose cohorts of 20, 40, 80 and 120 mg once daily, and two doses of Ad-RTS-hIL-12 (2x10^11vp and 1x10^12vp). Dose cohorts were treated at 10, 20, 30 and 40 mg of V. Only one dose of Ad-RTS-hIL-12 was explored (2x10^11vp). If ≥ 33% of subjects in the expansion cohort experience DLTs, additional subjects may be enrolled at the next lower dose, or at an intermediate dose, as recommended by the SRC. Grp 1: After 20mg cohort, SRC approved 40mg, which was deemed the MAD due to DLTs. SRC approved 30mg cohort to determine MTD, but due to poor compliance, SRC opened a 20mg exp cohort and then an intermediate 10mg cohort. Based on V compliance and efficacy, 20mg was determined to be the optimal dose

3. Secondary Outcome: Veledimex Pharmacokinetic Profile and Veledimex Concentration Ratio Between the Brain Tumor and the Blood
Description: From the protocol: Veledimex PK parameters to be determined will include, but are not limited to, the maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax), half-life (t1/2), area-under-the-concentration versus time curve (AUC), volume of distribution (Vd), and clearance (CL).
  From the SAP: The PK blood sample collection was performed either pre-dose or 3-5 hours post-dose, therefore only Cmax and Ctrough will be summarized and plotted. Veledimex concentration ratio between brain tumor and blood will be assessed on Day 0 samples. There will be no parameters including time to maximum plasma concentration (Tmax), half-life (t1/2), area under the curve (AUC), volume of distribution (Vd), and clearance (CL). Cmax will be determined from the maximum plasma concentration from Day 0 (post veledimex and resection/craniotomy), 3-5 hours after the veledimex dose on Day 1, and 3-5 hours after the veledimex dose on Day 14.
Time Frame: 15 days
Population: The Pharmacokinetic Population (PKP) includes all subjects who received veledimex and have PK samples to be measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 6 | 15 | 4 | 6 | 7
ng/mL
  Veledimex Plasma Cmax | 16.27 (8.68) | 41.77 (54.50) | 87.5 (35.86) | 52.76 (47.12) | 39.43 (35.18)
  Veledimex Plasma Ctrough | 3.60 (0.95) | 5.49 (2.57) | 11.72 (2.67) | 23.42 (15.51) | 4.39 (4.77)
  Veledimex metabolite: RG-116041 Plasma Cmax | 4.50 (2.38) | 8.57 (10.88) | 16.27 (9.39) | 10.17 (7.68) | 8.58 (5.96)
  Veledimex metabolite: RG-116041 Plasma Ctrough | 0.16 (0.19) | 0.50 (0.73) | 0.45 (0.79) | 2.44 (1.39) | 0.14 (0.24)
  Veledimex metabolite: RG-116043 Plasma Cmax | 0.83 (1.31) | 1.55 (2.11) | 3.62 (1.76) | 3.52 (2.80) | 1.93 (2.78)
  Veledimex metabolite: RG-116043 Plasma Ctrough | 0 (0) | 0.05 (0.18) | 0 (0) | 0.26 (0.37) | 0.06 (0.15)

4. Secondary Outcome: Cellular and Humoral Immune Responses Elicited by Ad-RTS-hIL-12 and Veledimex
Description: Peak serum IL-12 and I downstream IFN-gamma expressions between Day 3 to Day 28 are reported by dose cohort.
Time Frame: 28 days
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is denoted as the Per Protocol population in this uncontrolled setting.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 6 | 15 | 4 | 6 | 7
pg/mL
  Peak serum IL-12 | 51.2 (31.3) | 25.8 (7.1) | 65.7 (45.5) | 108.8 (41.0) | 25.1 (7.2)
  Peak serum IFN-gamma | 14.6 (7.1) | 57.0 (26.5) | 57.3 (46.5) | 125.5 (60.4) | 69.8 (48.8)

5. Secondary Outcome: Tumor Objective Response Rate (ORR)
Description: For the ORR calculation, responders are defined as those experiencing a confirmed complete response or confirmed partial response. Non-responders are those either with stable or progressive disease. Those subjects that cannot be assessed will be treated as non-responders for the purposes of deriving the percentage of responders and confidence intervals. The ORR is reported overall by treatment arm based on the investigator response at timepoints 56 days, Week 16, Week 24, and Week 48.
Time Frame: 48 weeks
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is to be used for analysis of dose limiting toxicities, overall survival and progression free survival and finding the maximum tolerated dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 6 | 15 | 4 | 6 | 7
Participants
  Complete Response | 0 | 1 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 1 | 0
  Stable Disease | 3 | 10 | 1 | 3 | 4
  Progressive Disease | 2 | 4 | 1 | 2 | 1
  Not Evaluable | 0 | 0 | 1 | 0 | 0
  No Response | 0 | 0 | 1 | 0 | 2
  Missing | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS (progression free survival) is the time in months from the first treatment (either veledimex or Ad-RTS-hIL-12) to the first assessment on which the overall response is reported as disease progression. Subjects withdrawing from the study will be censored at their last non progressive disease response assessment. If a subject does not have a non-progressive disease response assessment, the subject will be censored on the date of the first treatment as described above.
Time Frame: 3 years
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration.
Measure: Median (Full Range); unit: Months
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 4 | 15 | 4 | 6 | 4
Months | 4 [0.5 to 6] | 2 [0.5 to 12] | 0.25 [0 to 1] | 1.5 [0.5 to 24] | 1.75 [1 to 24]

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from the first dose of study drug (Day 0) to the date of death from any cause in days or months. Subjects are censored based on the last date known to be alive. For example:
  * Subjects who discontinue the study without documentation of additional follow-up will be censored at the date of discontinuation.
  * Subjects who are lost to follow-up will be censored at last follow-up contact date.
  * Subjects still alive up to 2 years from the first dose of study drug are classified as censored and as having completed all follow-up scheduling.
Time Frame: 6, 9, 12, 15, 18, and 24 months
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. Overall survival was reported by time point for the following set of subjects of the ESP: ATI001-102 Main Group 1: Craniotomy (treated at 20 mg veledimex: n=15).
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 0 | 15 | 0 | 0 | 0
percentage of participants
  Month 6 |  | 73.3 |  |  |
  Month 9 |  | 66.7 |  |  |
  Month 12 |  | 60.0 |  |  |
  Month 15 |  | 40.0 |  |  |
  Month 18 |  | 26.7 |  |  |
  Month 24 |  | 6.7 |  |  |

8. Secondary Outcome: Veledimex Concentration Ratio Between the Brain Tumor and the Blood
Description: as for outcome 3
Time Frame: 15 days
Population: The Pharmacokinetic Population (PKP) includes all subjects who received veledimex and have PK samples to be measured.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
Number analyzed (Participants) | 6 | 15 | 4 | 6 | 7
ratio | 0.42 (0.21) | 0.35 (0.30) | 0.51 (0.00) | 0.60 (0.33) | 0.63 (0.54)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Evaluation will be based on the incidence, intensity, and type of Adverse Events (AEs). Clinically significant changes in the subjects' physical examinations, vital signs, and ECG evaluations, and clinical manifestations relevant to abnormal laboratory values will be captured as AEs.
Arm/Group | Group 1 (Intracranial) 10 mg/Day Veledimex | Group 1 (Intracranial) 20 mg/Day Veledimex | Group 1 (Intracranial) 30 mg/Day Veledimex | Group 1 (Intracranial) 40 mg/Day Veledimex | Group 2 (Stereotactic) 20 mg/Day Veledimex
All-Cause Mortality (participants affected / at risk) | 6/6 | 12/16 | 4/4 | 5/6 | 5/7
Serious Adverse Events (participants affected / at risk) | 2/6 | 10/16 | 3/4 | 4/6 | 4/7
Other Adverse Events (participants affected / at risk) | 6/6 | 16/16 | 4/4 | 5/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Intracranial) 10 mg/Day Veledimex (N=6) | Group 1 (Intracranial) 20 mg/Day Veledimex (N=16) | Group 1 (Intracranial) 30 mg/Day Veledimex (N=4) | Group 1 (Intracranial) 40 mg/Day Veledimex (N=6) | Group 2 (Stereotactic) 20 mg/Day Veledimex (N=7)
Siezure (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain Oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural Hygroma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis Aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Intracranial) 10 mg/Day Veledimex (N=6) | Group 1 (Intracranial) 20 mg/Day Veledimex (N=16) | Group 1 (Intracranial) 30 mg/Day Veledimex (N=4) | Group 1 (Intracranial) 40 mg/Day Veledimex (N=6) | Group 2 (Stereotactic) 20 mg/Day Veledimex (N=7)
Headache (Nervous system disorders) | 4 (5) | 8 (12) | 1 (1) | 4 (5) | 3 (4)
Brain Oedema (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (2) | 1 (2)
Aphasia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive DIsorder (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Subdural Hygroma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemianopia Homonymous (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurologic Neglect Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reflexes Abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech Disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Field Defect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 8 (11) | 3 (5) | 3 (3) | 7 (8)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 4 (5) | 5 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (7) | 1 (1) | 3 (3) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 6 (7) | 4 (6) | 3 (5) | 1 (4)
Fatigue (General disorders) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 3 (4) | 0 (0) | 4 (8) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 2 (3) | 1 (1) | 3 (5) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (2)
Neutrophil Count Decreased (Investigations) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Amylase Increased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
C-Reactive Protein Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Liver Function Test Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Magnesium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Systolic Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein Total Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 4 (8) | 0 (0) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound Secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (3) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Communication Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor Retardation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 1 (3) | 2 (8) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (6) | 2 (2) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fluctuance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital Oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered Visual Depth Perception (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound Drainage (Surgical and medical procedures) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Incisional Drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Steroid Withdrawal Syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure shall not occur until (i) twenty-four (24) months have elapsed since Sponsor has notified Institution of the completion of the multi-center Study in order for Sponsor to comply with its obligations under 21 CFR 312.53(c)(4), or (ii) after the publication of the multi-center Study data, if the Study is a multi-center Study or Sponsor confirms in writing there will be no multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02026271/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT02026271/SAP_001.pdf